CLINICAL TRIAL: NCT01330407
Title: Comparative Assessment of Adjuvant Effect of Cultured Epidermal Autografts Versus Skin Allografts on Wound Healing of Burns Treated With Widely Expanded Skin Autograft Using Meek Micrografting Technique MEEKADEAU
Acronym: MEEKADEAU
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2009-A01247-50; 2009-31 (Other: AP HM)
Record Dates: First submitted 2011-04-05; First posted 2011-04-07 (Estimated); Last update posted 2015-11-20 (Estimated); Status verified 2015-11

CONDITIONS: Burn Wounds
MeSH Terms: conditions — Burns

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- gp2 (Experimental): Cultured Epidermal Autografts
  Interventions: Procedure: Cultured Epidermal Autografts
- gp1 (Active Comparator): cryopreserved skin allografts.
  Interventions: Procedure: cryopreserved skin allografts.

INTERVENTIONS:
Procedure: cryopreserved skin allografts.
  Arms: gp1
Procedure: Cultured Epidermal Autografts
  Arms: gp2

SUMMARY:
The investigators intend to conduct a comparative, monocentric prospective double-blind study with intra-subject randomization, to compare the results on wound healing of 2 adjuvant treatments to Meek micrografting technique : Cultured Epidermal Autografts and cryopreserved skin allografts.

DETAILED DESCRIPTION:
10 patients presenting burn wounds over 50% of total body surface area, including at least 40 % of deep burns, will be enrolled.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females between 18 to 60 years of age
2. Burns > 50% Total Body Surface Area (TBSA), including deep burns > 40% TBSA (deep partial thickness and full thickness burns).
3. Patients presenting two 300 cm² (30x10cm) non adjacent burn wound areas, of similar depth assessed by Laser Doppler Imaging, on body anterior side, functional areas excepted.
4. Written informed consent, signed by patient or legal representative (if patient unable to sign).
5. Negative pregnancy test

Exclusion Criteria:

1. Chemical or electric burns
2. Short delay life threatening disease, by itself or when associated with burns.
3. Chronic systemic steroïd intake,
4. Pre-existing diseases interfering with wound healing : inherited connective tissue disorder (Ehlers Danlos syndrome, Marfan syndrome), Epidermolysis Bullosa. Medical treatment interfering with wound healing (retinoids..).
5. Prisonners
6. Pregnant women
7. Patient under guardianship.
8. Participation in another investigational trial within this trial

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Estimated)
Dates: Start 2011-04; Primary Completion 2016-03 (Estimated); Study Completion 2016-03 (Estimated)

PRIMARY OUTCOMES:
TIME OF HEALING | 2 YEARS
  to compare wound healing speed on the 2 treated areas, considering epithelialization rate until complete wound healing.

SECONDARY OUTCOMES:
QUALITY OF HEALING | 2 YEARS
  to assess the quality of wound healing and scar maturation.

CONTACTS AND LOCATIONS:
Overall Officials: BERNARD BELAIGUES, Study Director — Assistance Publique hôpitaux de Marseille
Locations (1):
- Assistance Publique Hopitaux de Marseille, Marseille, France